CLINICAL TRIAL: NCT00548652
Title: Role of Apathy in the Effectiveness of Weight Loss Interventions in Obese Patients
Brief Title: Role of Apathy in the Effectiveness of Weight Loss Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Nebraska Western Iowa Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Prasad R. Padala, Staff Physician, VA Nebraska Western Iowa Health Care System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00469
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Obesity; Apathy
Keywords: apathy; obesity; methylphenidate; MOVE; medical crisis counselling
MeSH Terms: conditions — Obesity; Lethargy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (No Intervention): standard nutrition counselling
- 2 (Experimental): MOVE -weight loss intervention
  Interventions: Behavioral: MOVE
- 3 (Experimental): MOVE plus medical crisis counselling
  Interventions: Behavioral: medical crisis councelling; Behavioral: MOVE
- 4 (Experimental): MOVE plus methylphenidate
  Interventions: Drug: methyphenidate; Behavioral: MOVE
- 5 (Experimental): MOVE plus methyphenidate plus medical crisis counselling
  Interventions: Drug: methyphenidate; Behavioral: medical crisis councelling; Behavioral: MOVE

INTERVENTIONS:
Behavioral: MOVE — is a VA based multidesciplinary weight loss intervention
  Arms: 2
Behavioral: medical crisis councelling — group counselling sessions
  Arms: 3
Behavioral: MOVE — is a VA based multidesciplinary weight loss intervention
  Arms: 3
Drug: methyphenidate — methyphenidate will be used to treat apathy dose 10mg bid
  Arms: 4
Behavioral: MOVE — is a VA based multidesciplinary weight loss intervention
  Arms: 4
Drug: methyphenidate — methyphenidate will be used to treat apathy dose 10mg bid
  Arms: 5
Behavioral: medical crisis councelling — group counselling sessions
  Arms: 5
Behavioral: MOVE — is a VA based multidesciplinary weight loss intervention
  Arms: 5

SUMMARY:
The purpose of this study is to determine whether treating apathy with methylphenidate or medical Crisis counselling will increase adherence to weight loss programs thereby increasing their effectiveness

DETAILED DESCRIPTION:
Title: The role of Apathy in the effectiveness of weight loss interventions in obese patients

Objective: Obesity is a major public health problem. Apathy is a common behavioral problem characterized by loss of initiative, poor motivation and persistence. Presence of apathy impairs the self-care behavior in obese patients. Lack of novelty might impair a patient's ability to seek new interactions, life styles and new treatment options for obesity. Lack of motivation might impair a patient's ability to initiate exercise regimen or diet whereas lack of persistence impairs the compliance with these regimens. Thus, apathy influences all stages of self-care. We hypothesize that the treatment of apathy will result in better adherence to weight loss interventions in obese veterans enrolled in the MOVE program.

Research Design: A prospective open label randomized study. Group 1 will have patients with obesity as defined as BMI>30, and apathy defined as AES score of > 40. This group will be treated with standard nutrition counseling. Group 2 will have patients with obesity and apathy as defined above and will receive the MOVE enhancement program alone (The MOVE program is a national VA weight loss program). Group 3 will be treated with methylphenidate along with the MOVE enhancement program. Group 4 will be treated with medical crisis counseling along with the MOVE enhancement program. Group 5 will be treated with methylphenidate, and the medical crisis counseling along with the MOVE enhancement program.

Methodology: 30 patients meeting the criteria will be enrolled in each of the five arms. All patients will be in the study for duration of six months. All patients in the methylphenidate arm will be started at 5mg twice daily and titrated to 10mg twice daily at two weeks. Patients will be assessed on regular intervals using the Apathy Evaluation Scale, Hamilton Depression Scale and the Patient activation measure. MOVE sessions will be held once weekly from the 2nd visit to the end of the study. Medical Crisis Counseling visits will be every week for nine sessions and then every other week till the end of the study

Clinical Relationships/Significance: The prevalence of obesity in the general population is over 30%. However the prevalence of obesity in the VA health system is almost 70%. Since obesity predisposes to several co-morbid conditions such as hypertension, diabetes and cardiovascular disease, it is important to develop interventions that are effective in inducing weight loss. Since apathy plays a large role in the self care behaviours that lead to obesity, treating apathy may improve adherence to weight loss programs

ELIGIBILITY:
Inclusion Criteria:

* BMI >30
* Apathy score >40

Exclusion Criteria:

* History of cancer, except basal cell
* Cardiovascular event in last 6 months
* Renal failure

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2007-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cyrus DeSouza, MD, Principal Investigator — VA Medical Center, Omaha
Locations (1):
- VA Medical Center, Omaha, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: standard nutrition counselling
- VA MOVE: MOVE -weight loss intervention
  MOVE: is a VA based multidesciplinary weight loss intervention
- Intervention: MOVE plus methylphenidate
  methyphenidate: methyphenidate will be used to treat apathy dose 10mg bid
  MOVE: is a VA based multidesciplinary weight loss intervention
Period: Overall Study
Arm/Group | Usual Care | VA MOVE | Intervention
Started | 18 | 38 | 45
Completed | 16 | 29 | 34
Not Completed | 2 | 9 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | VA MOVE | Intervention | Total
Number analyzed (Participants) | 18 | 38 | 45 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (14.3) | 55.2 (10.1) | 52.5 (10.4) | 52.34 (10.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16 | 32
  Male | 9 | 31 | 29 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 4 | 3 | 7 | 14
  White | 12 | 32 | 38 | 82
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 38 | 45 | 101
BMI [Mean (Standard Deviation); unit: kg/m^2] | 36.06 (5.91) | 38.78 (5.6) | 37.58 (5.69) | 37.21 (5.55)
Apathy Evaluation Scale [Mean (Standard Deviation); unit: units on a scale] — Score range 18-72 Higher score indicates more apathy
  units on a scale | 41.89 (8.2) | 42.12 (7.93) | 42.96 (8.94) | 42.06 (7.94)

OUTCOME MEASURES:

1. Primary Outcome: Apathy Evaluation Scale
Description: Apathy Evaluation Scale (AES) measures apathy over the previous four weeks Scale range: 18 (minimum score)- 72 (Maximum score) Higher scores indicate higher apathy Better outcome would be reduction in the score
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | VA MOVE | Intervention
Number analyzed (Participants) | 16 | 29 | 34
units on a scale | -7.69 (6.77) | -6.4 (7.35) | -6.15 (8.3)

2. Secondary Outcome: Change in Weight
Description: value at 6 months minus value at baseline
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Usual Care | VA MOVE | Intervention
Number analyzed (Participants) | 16 | 29 | 34
Kg | -0.6 (3.73) | -0.61 (7.14) | -4.61 (9.42)

ADVERSE EVENTS:
Arm/Group | Usual Care | VA MOVE | Intervention
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/38 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/38 | 0/45
Other Adverse Events (participants affected / at risk) | 0/18 | 0/38 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes